CLINICAL TRIAL: NCT04727489
Title: Study of the Genetic Factors Involved in Autism and Related Disorders
Acronym: Gene&autism
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-89
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; developmental Disorder; gene; polymorphism; mutation
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from subjects will be stored in the biobank of our study. From some patients with deleterious mutations in synaptic genes,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Autism Spectrum Disorder: Probands with Autism Spectrum Disorder, (N=700), Diagnosis of ASD according to DSM-V criteria For all patients included in the study, core assessment carried out by either collaborating partners consists of diagnosis using the Autism Diagnostic Interview-Revised (ADI-R) criteria for autism and Autism Diagnostic Observation Schedule (ADOS-G) criteria for autism or Autism Spectrum Disorders. Patients with profound intellectual disability or with a known medical cause of autism, such as neurocutaneous syndromes, Fragile X, metabolic disorders, extreme prematurity, congenital rubella and other prenatal or postnatal neurological infections or gross dysmorphology, will be excluded.
  Interventions: Genetic: DNA from subjects will be stored in the biobank of our study.
- Control without Autism Spectrum Disorder: Controls without Austim Spectrum Disorder, aged 6 to 40, N=2100 (300 adultes, 300 children) Healthy individuals with or without idiopathic surgical or urological conditions (e.g. orthopaedic conditions, hernia repairs, renal malformations, pre- or post-circumcision, phimosis, balanitis, scoliosis, congenital hip dislocation, adenoid or tonsil removal, dental procedures such as wisdom tooth extraction, cosmetic procedures such as removal of skin tags or cleft lip repairs, non-head injuries such as fractures, drainage of subungual or perichondrial haematomata).
  Interventions: Genetic: DNA from subjects will be stored in the biobank of our study.
- Relatives of probands with Autism Spectrum Disorder: Relatives of probands with Autism Spectrum Disorder (N=1200 parents, N=600 siblings, N=300 other relatives)
  * Without Autism Spectrum Disorder diagnosis according to DSM-V,
  * With Autism Spectrum Disorder diagnosis according to DSM-V, and using the Autism Diagnostic Interview-Revised (ADI-R) criteria for autism and Autism Diagnostic Observation Schedule (ADOS-G) criteria for autism or Autism Spectrum Disorders
  Interventions: Genetic: DNA from subjects will be stored in the biobank of our study.
- Relatives of controls: Relatives of controls without Autism Spectrum Disorder, N=400 first degree relatives
  Interventions: Genetic: DNA from subjects will be stored in the biobank of our study.

INTERVENTIONS:
Genetic: DNA from subjects will be stored in the biobank of our study. — Diagnostic Interview-Revised (ADI-R) criteria for autism and Autism Diagnostic Observation Schedule (ADOS-G) criteria for autism or Autism Spectrum Disorders.
  Other Names: diagnostic test

SUMMARY:
The main objective of the study is to define, for Autism Spectrum Disorder, the extent of genetic variation in synaptic pathways that may be targeted for therapeutic development. For this purpose the investigators will take advantage of large, well-characterized cohorts of patients with Autism Spectrum Disorder for genetic screenings. Targeted sequencing of selected synaptic genes, previously associated with Autism Spectrum Disorder, will be carried out in these cohorts with deep coverage of coding regions and a strong focus on previously untested regulatory regions. Genomic data from Copy Number Variant, whole genome sequencing and exome sequencing, available for some of these patients, will be integrated in the overall analysis. The investigators will strongly emphasize the establishment of comprehensive genotype/phenotype correlations.

DETAILED DESCRIPTION:
Aim 1: To identify genetic variants in selected synaptic genes, by targeted sequencing with deep coverage of coding regions and a strong focus on previously untested regulatory regions in Autism Spectrum Disorder

Aim 2: To define the range of clinical phenotypes caused by mutations in synaptic genes by establishing detailed genotype/phenotype correlations and analyzing segregation in families with multiple individuals affected by Autism Spectrum Disorder, Autism Spectrum Disorder traits or other neuropsychiatric disorders

Aim 3: To identify the neuronal phenotypes caused by deleterious synaptic mutations for further translational studies

ELIGIBILITY:
Inclusion Criteria---------------------------------------------------------------------------------------------------

Probands with Autism Spectrum Disorder

* Meet the diagnostic criteria for ASD of the DSM-5 [American Psychiatric Association, 2013] based on a consensus between the clinical expertise of expert clinicians, the scores of the Autism Diagnostic Interview-Revised (ADI-R) (Rutter et al, 2003) and those of the Autism Diagnosis Observation Schedule (ADOS-2) (Lord et al, 2012)
* Be at least 24 months (no upper age limit)
* Somatic and Intellectual state compatible with a blood test
* Affiliation to the social insurance
* Signature of informed consent by the applicant or by holders of parental authority if the subject is a minor or by the guardian if the subject is under guardianship

Controls without ASD

* At least 24 months old
* Somatic and Intellectual state compatible with a blood test
* Affiliation to the social insurance
* Signature of informed consent by the subject or by holders of parental authority if the subject is a minor or by the guardian if the subject is under guardianship

Relatives of the probands with ASD or of controls without ASD

* At least 24 months old
* Somatic and Intellectual state compatible with a blood test
* Affiliation to the social insurance
* Signature of informed consent by the subject or by holders of parental authority if the subject is a minor or by the guardian if the subject is under guardianship

Exclusion Criteria --------------------------------------------------------------------------------------------------

Probands with Autism Spectrum Disorder

* Severe Intelectual Deficiency (IQ,35 or developmental age <18 months)

  ●. Personal psychiatric history (schizophrenia, bipolar disorder, substance use disorder (except tobacco), recurrent depression disorder, severe instable anxiety disorder)
* Personal neurologic history (epilepsy, or severe neurological disease)

Relatives of the probands with ASD, of the controls or the controls:

● Medical condition (psychiatric or somatic) not compatible with the inclusion

Ages: 24 Months to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For all patients included in the study
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2036-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of synaptic gene deleterious mutations in patients with Autism Spectrum Disorder | up to 12 months after completion of the inclusion and molecular explorations
  Prevalence of synaptic gene deleterious mutations in patients with Autism Spectrum Disorder

SECONDARY OUTCOMES:
Prevalence of the deleterious mutations in the major biological pathways in Autism Spectrum Disorder | up to 12 months after completion of the inclusion and molecular explorations
  The deleterious mutations that the investigators will identify in genes related to Autism Spectrum Disorders will help to have a comprehensive framework of biological pathways involved in Autism Spectrum Disorder

CONTACTS AND LOCATIONS:
Overall Officials: Richard Delorme, M.D, Ph.D, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (6):
- France (6):
  - Centre de rehabilitation psychosociale, Hopital Saint Egreve, Grenoble, Grenoble
  - CIC, CHU Bordeaux, Bordeaux
  - CRA, Hopital Charles Perrens, Bordeaux, Bordeaux
  - CIC, H. Mondor, Creteil, Créteil
  - Albert Chenevier Hospital, Créteil, Île-de-France Region
  - Robert Debré Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delorme R, Ey E, Toro R, Leboyer M, Gillberg C, Bourgeron T. Progress toward treatments for synaptic defects in autism. Nat Med. 2013 Jun;19(6):685-94. doi: 10.1038/nm.3193. Epub 2013 Jun 6. PMID 23744158
- See also: Description website of the sponsor — http://www.inserm.fr
- Available data/document: Study Protocol — http://www.inserm.fr
- Available data/document: Informed Consent Form — http://www.inserm.fr